CLINICAL TRIAL: NCT02941341
Title: Ambispective Observational Post-Authorisation Study on the Use of Bemfola® in Human Assisted Reproductive Techniques in Spain.
Brief Title: Observational Post-Authorisation Study on the Use of Bemfola® in Human Assisted Reproductive Techniques in Spain.
Acronym: BIRTH
Status: Completed | Type: Observational
Sponsor: Finox AG (Industry)
Responsible Party: Sponsor
Other Study IDs: FIN-BEM-2015-01
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Infertility
Keywords: Bemfola; r-hFSH; ART; Oocytes; OHSS; Pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: r-hFSH — As per standard practice
  Other Names: Bemfola

SUMMARY:
Non-comparative, observational, ambispective post-authorisation study (EPA-SP).

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Currently undergoing an IVF or ICSI cycle or are oocyte-donors
* Have completed controlled ovarian stimulation
* Have received at least 5 doses of Bemfola®
* Are pituitary suppressed with a GnRH antagonist
* Have undergone oocyte retrieval
* Have signed the Informed Consent Form

Exclusion Criteria:

* Hypersensitivity to the active substance follitropin alfa, FSH or to any of the excipients listed
* Presence of tumours of the hypothalamus or pituitary gland

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have undergone oocyte retrieval after ovarian stimulation with Bemfola®, either as part of an in vitro fertilisation (IVF) cycle or with an intracytoplasmic sperm injection (ICSI), for reproductive purposes or for oocyte donation, and who are pituitary-suppressed with a GnRH antagonist.
Sampling Method: Non-Probability Sample
Enrollment: 1222 (Actual)
Dates: Start 2016-10; Primary Completion 2018-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Total number of oocytes retrieved | 34-36 hours after hCG administration and after a maximum 16 days of r-hFSH treatment

SECONDARY OUTCOMES:
Number of fertilised oocytes | 1 day after ovum pick-up
Quality of oocytes | At Day 4-5
Number and quality of transferred embryos | Day of embryo transfer, either 2,3 or 5 days after oocyte retrieval
Fertilization and implantation rate | 5 to 6 weeks after oocyte retrieval
Incidence of serious adverse events, including moderate-to-severe OHSS | From Day 1 of stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Ferrando, MD, Principal Investigator — Director IVI Bilbao, Spain; Buenaventura Coroleu Lletget, MD, Principal Investigator — Jefe del Servicio de Medicina de la Reproducción,Hospital Universitari Quirón Dexeus, Barcelona, Spain; Luis Rodríguez-Tabernero Martín, MD, Principal Investigator — Jefe de la Unidad de Reproducción, Hospital Clínico Universitario de Valladolid, Valladolid, Spai^n
Locations (1):
- IVI Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferrando M, Coroleu B, Rodriguez-Tabernero L, Barrenetxea G, Guix C, Sanchez F, Jenkins J; BIRTH study group. The continuum of ovarian response leading to BIRTH, a real world study of ART in Spain. Fertil Res Pract. 2020 Jul 29;6:13. doi: 10.1186/s40738-020-00081-4. eCollection 2020. PMID 32742711